CLINICAL TRIAL: NCT07228741
Title: Resistance Exercise and Incretin Mimetic for Cardiometabolic Health in Survivors of ALL With Obesity
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESIST; NCI-2026-00106 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2025-11-10; First posted 2025-11-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Acute Lymphoblastic Leukemia; Obesity
Keywords: ALL; ALL Survivors
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Obesity | interventions — Tirzepatide; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adult survivors of childhood acute lymphoblastic leukemia (ALL) (Experimental): This is a 28-week, single-arm, open-label phase II clinical trial evaluating the combination of Tirzepatide and remote, supervised, tailored resistance exercise training to achieve weight loss in adult survivors of childhood acute lymphoblastic leukemia (ALL) living with obesity or overweight with comorbidity. The primary goal is to achieve ≥5% weight loss while preserving lean muscle mass.
  Interventions:
  * Tirzepatide: Weekly subcutaneous injections starting at 2.5 mg, titrated every 4 weeks up to 15 mg as tolerated.
  * Resistance Exercise: Remote, supervised, tailored resistance training 3 times per week for 28 weeks.
  * Lifestyle Counseling: Every 4 weeks focused on balanced diet and caloric deficit.
  Interventions: Drug: Tirzepatide; Behavioral: Resistance Exercise; Behavioral: Lifestyle Counseling

INTERVENTIONS:
Drug: Tirzepatide — A once-weekly subcutaneous injection starting at 2.5 mg and dose escalation every 4 weeks up to a maximum of 15 mg, following FDA-approved guidelines. Dose escalation may be paused for exceptional responders.
Behavioral: Resistance Exercise — A remote, supervised, tailored program delivered via a digital platform, with three sessions per week. Supervision is reduced over time (initially 2x/week, then reduced gradually).
Behavioral: Lifestyle Counseling — Provided every 4 weeks, focusing on balanced diet, caloric deficit, and symptom management.

SUMMARY:
This is a 28-week, single-arm, open-label phase II clinical trial evaluating the combination of Tirzepatide and remote, supervised, tailored resistance exercise training to achieve weight loss in adult survivors of childhood acute lymphoblastic leukemia (ALL) living with obesity or overweight with comorbidity.

Primary Objective(s):

• To evaluate the effectiveness for weight loss of the combined intervention using once weekly Tirzepatide plus remote, supervised, tailored resistance exercise (three sessions per week) in adult survivors of childhood ALL with obesity or overweight (BMI ≥27 kg/m2) with ≥1 weight-related comorbidity (hypertension, dyslipidemia, obstructive sleep apnea, or cardiovascular disease). The effectiveness will be estimated as the proportion of evaluable participants who achieve at least 5% weight loss from baseline to week 28.

The study will target a proportion of participants achieving 5% weight loss of 70% and consider fewer than 40% achieving 5% weight loss as unacceptable.

Secondary Objective(s):

* Estimate the proportion of participants who adhere to the 28-week combined intervention. Adherence to Tirzepatide will be defined as receiving at least 70% of prescribed doses. Adherence to resistance exercise will be defined as attending at least 50% of prescribed exercise sessions. Adherence to the combined intervention will be considered if participants complete the study and meet both the Tirzepatide and exercise adherence endpoint. The adherence to each component of the intervention will also be reported.
* Estimate the average percentage weight loss from week 0 to 28 for participants completing the combined 28-week intervention. The study will target a mean weight reduction of 10% and consider <5% unacceptable.

DETAILED DESCRIPTION:
Survivors of childhood ALL are at increased risk for obesity and cardiometabolic disease. Tirzepatide is FDA-approved for weight management in adults and results in significant weight loss but may cause lean mass loss. Resistance exercise programs are feasible and effective in this population.

This study evaluates the efficacy of combining Tirzepatide with resistance exercise in adult survivors of ALL treated with chemotherapy only and at least 2 years off therapy.

The primary objective is to estimate the proportion of participants achieving ≥5% weight loss over 28 weeks. Secondary objectives include adherence to the intervention and changes in body composition, cardiometabolic health, and aging biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* ≥5 years from diagnosis of acute lymphoblastic leukemia (ALL) treated with chemotherapy only
* ≥2 years from completion of therapy
* Participant has a negative (urine or blood) pregnancy test (if female)

Consistent with the FDA-approval for marketing of Tirzepatide for the treatment of obesity:

* Age ≥18 years at the time of enrollment
* Participant has obesity (BMI > 30kg/m2) or overweight (BMI > 27kg/m2) with ≥1 weight related co-morbidity (hypertension, dyslipidemia, obstructive sleep apnea, cardiovascular disease)

  * hypertension: treated or with systolic blood pressure (SBP) ≥130 mmHg or diastolic blood pressure (DBP) ≥80 mmHg
  * dyslipidemia: treated or with low-density lipoprotein (LDL) ≥160 mg/dL (4.1 mmol/L) or triglycerides ≥150 mg/dL (1.7 mmol/L), or high-density lipoprotein (HDL) <40 mg/dL (1.0 mmol/L) for men or HDL<50 mg/dL (1.3 mmol/L) for women
  * obstructive sleep apnea
  * cardiovascular disease (for example, ischemic cardiovascular disease, New York Heart Association (NYHA) Functional Class I-III heart failure)

Exclusion Criteria:

* Participant has known diabetes or is found at baseline to have laboratory evidence of diabetes including HbA1c ≥ 6.5%
* Participant is using or has used weight management medication in the past 3 months or had recent significant weight loss > 5kg in the last 3 months Severe renal dysfunction (eGFR <30 mL/min/1.73 m²)

  * Saxenda® (liraglutide 3.0 mg)
  * Xenical®/Alli® (orlistat)
  * Meridia® (sibutramine)
  * Acutrim® (phenylpropanolamine)
  * Sanorex® (mazindol)
  * Adipex® (phentermine)
  * BELVIQ® (lorcaserin)
  * Qsymia® (phentermine/topiramate combination)
  * Contrave® (naltrexone/bupropion)
  * Compounded or generic incretin mimetic (GLP-1) medication

Note: Use of metformin or any other glucose-lowering medication, whether prescribed for polycystic ovary syndrome or diabetes prevention is not permitted.

* Participant has Multiple Endocrine Neoplasia Type 2 (MEN2) or family history of medullary thyroid cancer
* Participant has severe renal dysfunction (renal-eGFR <30 mL/min/1.73)
* Participant has history of major cardiovascular event in past 3 months (e.g. acute myocardial infarction, cerebrovascular accident, unstable angina, hospitalization due to congestive heart failure or currently NYHA class IV heart failure symptoms)
* Participant has uncontrolled hypertension during clinic assessment (SBP ≥160 mmHg or DBP ≥100 mmHg) ▪ Participant has known acute or chronic hepatitis or signs and symptoms of other liver disease determined by alanine aminotransferase test (ALT) > 3 times the upper normal limit
* Participant has known chronic pancreatitis or recent acute pancreatitis (in the past 1 year)
* Participant is pregnant, or within 3 months post-partum, or nursing, or planning to become pregnant
* Participant has clinically significant gastric emptying abnormality or chronically takes medications that affect GI motility (does not include Proton pump inhibitor (PPI) or histamine 2 blockade)
* Participant has a transplanted organ or awaiting a transplant
* Participant has current active cancer or undergoing treatment for active cancer
* Participant has untreated hypothyroidism with thyroid-stimulating hormone (TSH) > 10 uIU/mL or symptomatic
* Participant has severe mental health disorder (e.g.major depressive disorder, schizophrenia, bipolar disorder, or other serious mood or anxiety disorder) or a history of suicide attempt
* Participant has a patient health questionnaire-8 (PHQ-8) score of 15 or more at screening
* Participant has a history of known drug or alcohol use disorder that in the opinion of the investigator may preclude the participant from following and completing the protocol
* Participant has history of self-reported marijuana use in the past 3 months and unwilling to abstain during the trial.
* Participant is unwilling or unable to perform self-injections of study drug (visually impaired or physically limited) and does not have assistance of a sighted individual/support person who is trained
* Participant has cognitive impairment that, in the opinion of the investigator, would preclude the ability to participate in the intervention including self-injections and virtual study visits
* Participant is Non-English speaking
* Participant has no access to a smartphone with Bluetooth for accelerometer and WiFi availability for exercise sessions
* Participant lives in a state that we cannot ship medication per current St. Jude Pharmacy restrictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness for weight loss of the combined intervention using once weekly Tirzepatide plus remote, supervised, tailored resistance exercise. | 28 weeks (assessed baseline and Week 28)
  The effectiveness will be estimated as the proportion of evaluable participants (those completing both week 0 and 28 visits) who achieve at least 5% weight loss from baseline to week 28.

SECONDARY OUTCOMES:
To estimate the proportion of participants who adhere to the 28-week combined intervention. | 28 weeks
  Adherence to Tirzepatide will be defined as receiving at least 70% of prescribed doses. Adherence to resistance exercise will be defined as attending at least 50% of prescribed exercise sessions. Adherence to the combined intervention will be considered if participants complete the study and meet both the Tirzepatide and exercise adherence endpoint.
To estimate the average percentage weight loss from week 0 to 28 for participants completing the combined 28-week intervention. | 28 weeks
  Weight will be monitored at each visit to determine the total amount of weight loss from week 0 to week 28.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie B Dixon, MD, MPH, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols